CLINICAL TRIAL: NCT00003790
Title: Detection of Minimal Residual Disease in Children Receiving Therapy for AML or MDS
Brief Title: Detection of Residual Disease in Children Receiving Therapy for Acute Myeloid Leukemia or Myelodysplastic Syndrome
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: B942; CCG-B942 (Other: Children's Cancer Group); CDR0000066930 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2004-04-23 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: recurrent childhood acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — Polymerase Chain Reaction; Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: polymerase chain reaction
Other: flow cytometry

SUMMARY:
RATIONALE: Diagnostic procedures may improve the ability to detect residual disease.

PURPOSE: Clinical trial to detect the presence of residual disease in children who are receiving therapy for acute myeloid leukemia or myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the frequency and prognostic significance of persistent abnormal cells with an aberrant phenotype detected by multidimensional flow cytometry (MDF) in bone marrow samples from children who have achieved clinical remission after receiving treatment for acute myeloid leukemia or myelodysplastic syndrome. II. Compare the frequency of persistent abnormal cells obtained by MDF with that of polymerase chain reaction (PCR), morphologic, and cytogenetic analyses of these patient samples. III. Determine the frequency and prognostic significance of persistent abnormal cells with a leukemia-specific molecular marker detected by PCR in samples from these patients.

OUTLINE: Patients have bone marrow samples collected during the course of therapy on the CCG 2961 acute myeloid leukemia treatment protocol. These samples are collected: 1. At the time of diagnosis 2. At the end of induction (within a week of day 35) 3. At the end of consolidation (before bone marrow transplant or Capizzi 2) 4. Before and after interleukin-2 (IL-2) therapy, if applicable 5. At the end of therapy (after transplant with evidence of engraftment for autologous bone marrow transplant patients; after course 2 of intensification for chemotherapy patients; and after IL-2 day 21 for IL-2 patients) 6. At relapse, if applicable. The presence of minimal residual disease in bone marrow is assessed using multidimensional flow cytometry and PCR.

PROJECTED ACCRUAL: A total of 400 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Acute myeloid leukemia (AML) or myelodysplastic syndrome and enrolled on the CCG 2961 AML treatment protocol Must have one of the following cytogenetic abnormalities t(8;21) inv(16) abnormality of 11q23 OR All patients being enrolled for interleukin-2 therapy or standard care can be enrolled at the time of randomization

PATIENT CHARACTERISTICS: Age: Children Performance status: Specified on the CCG 2961 AML treatment protocol Life expectancy: Specified on the CCG 2961 AML treatment protocol Hematopoietic: Specified on the CCG 2961 AML treatment protocol Hepatic: Specified on the CCG 2961 AML treatment protocol Renal: Specified on the CCG 2961 AML treatment protocol

PRIOR CONCURRENT THERAPY: Specified on the CCG 2961 AML treatment protocols

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with acute myeloid leukemia or myelodysplastic syndrome (MDS) enrolled on the CCG 2961 AML treatment protocol.
Sampling Method: Non-Probability Sample
Enrollment: 496 (Actual)
Dates: Start 1995-02; Primary Completion 2002-04 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Determine the frequency and prognostic significance of persistent abnormal cells with an aberrant phenotype detected by MDF in bone marrow samples from patients who have achieved clinical remission. | 12 months from achievement of remission

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sievers, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (43):
- United States (40):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Children's Hospital of Denver, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Wayne Hughes Institute, Roseville, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Fargo, Fargo, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Center for Cancer Treatment and Research, Columbia, South Carolina
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Grace Health Centre, Halifax, Nova Scotia

REFERENCES:
- [Derived] Vujkovic M, Attiyeh EF, Ries RE, Goodman EK, Ding Y, Kavcic M, Alonzo TA, Wang YC, Gerbing RB, Sung L, Hirsch B, Raimondi S, Gamis AS, Meshinchi S, Aplenc R. Genomic architecture and treatment outcome in pediatric acute myeloid leukemia: a Children's Oncology Group report. Blood. 2017 Jun 8;129(23):3051-3058. doi: 10.1182/blood-2017-03-772384. Epub 2017 Apr 14. PMID 28411282